CLINICAL TRIAL: NCT02951741
Title: Relations Between Hematologic Variables and Postoperative Bleeding and Transfusion in Revision Total Hip Replacement Arthroplasty
Brief Title: Revision Total Hip Replacement Arthroplasty and Hematologic Variables
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Associate Professor, Seoul National University Bundang Hospital
Other Study IDs: B-1502/288-302
Record Dates: First submitted 2016-10-24; First posted 2016-11-01 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Avascular Necrosis of Hip; Degenerative Hip Joint Disease
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RTHRA group: patients undergoing revision total hip replacement
  Interventions: Other: RTHRA group

INTERVENTIONS:
Other: RTHRA group — hematologic variables measurement in patients undergoing revision total hip replacement

SUMMARY:
Revision total hip replacement arthroplasty is a surgery having intra- and postoperative substantial blood loss. The investigators will investigate the relationship between the various hematologic variables and postoperative bleeding volume.

ELIGIBILITY:
Inclusion Criteria:

* revision total hip replacement

Exclusion Criteria:

* hematologic disease
* anticoagulant medication
* American Society of Anesthesiologists physical status 4 and 5

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing revision total hip replacement
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change of FIBTEM | 5 minutes before initiation of anesthesia and 5 minutes after finishing operation
  FIBTEM: one of the measurements of the rotational thromboelastometry

SECONDARY OUTCOMES:
volume of infused fluid during operation | Period from starting to finishing the operation (During operation, an expected average of 3 hours)
  Infused total crystalloid and colloid volume during the operation will be recorded
intraoperative urine output | Period from starting to finishing the operation (During operation, an expected average of 3 hours)
transfusion units | Period from starting to finishing the operation (During operation, an expected average of 3 hours) and postoperative first day
  Red blood cell
postoperative bleeding volume | postoperative 72 hours
Hemoglobin | preoperative day 1
Hemoglobin | postoperative day 4
Hematocrit | preoperative day 1
Hematocrit | postoperative day 4
Platelet count | preoperative day 1
Platelet count | postoperative day 4
prothrombin time_international normalized ratio | preoperative day 1
prothrombin time_international normalized ratio | postoperative day 1
activated partial prothrombin time | preoperative day 1
activated partial prothrombin time | postoperative day 1
fibrinogen concentration | preoperative day 1
fibrinogen concentration | postoperative day 1

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Seok Na, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No